CLINICAL TRIAL: NCT00353067
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Examine the Safety and Efficacy of Veliflapon (DG-031) in Reducing the Risk of Acute Cardiovascular Events in African American Patients With Coronary Artery Disease(The LTCAD Study).
Brief Title: Veliflapon (DG-031)to Prevent Heart Attacks or Stroke in Patients With a History of Heart Attack or Unstable Angina
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: deCODE genetics (Industry)
Collaborators: Henry Ford Health System (Other); Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DG-031-CV-301
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Acute Coronary Syndrome
Keywords: unstable angina; myocardial infarction; coronary thrombosis; coronary atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Myocardial Infarction; Coronary Thrombosis; Coronary Artery Disease | interventions — 2-(4-(quinolin-2-yl-methoxy)phenyl)-2-cyclopentylacetic acid

INTERVENTIONS:
Drug: veliflapon (DG-031)

SUMMARY:
The purpose of this study is to determine if veliflapon (DG-031)can prevent a heart attack or stroke in African American patients with a history of unstable angina or myocardial infarction.

DETAILED DESCRIPTION:
Genetic linkage and association studies in Icelandic patients with a history of myocardial infarction and stroke showed common haplotypes in two genes, 5-lipoxygenase activating protein(FLAP)and Leukotriene A4 Hydrolase(LTA4H), that each conferred significant risk for MI and stroke. The FLAP haplotype had a RR of 1.8 for MI and 2.1 for those with MI and stroke. LTA4H haplotype had a RR of 1.1 for MI and 1.5 for MI and stroke.Both gene associations were replicated in European and US Caucasian groups and were independent of the conventional risk factors such as LDL-cholesterol, hypertension, and diabetes. The haplotype for the LTA4H pathway showed a modest relative risk of 1.2 in US Caucasian cohorts for all MI and 1.4 for MI and stroke. However, the LTA4H haplotype had a much higher relative risk of 3.5 for myocardial infarction in African-Americans (p=0.000022).

Self identified African American patients with acute coronary syndrome (ACS) were selected for this study as this population has the highest risk identified to date for developing an MI related to the HapK genetic variant in the leukotriene pathway. The study will be enriched to include African American patients randomized by an algorithm designed to assure that approximately 80% of the study population will be Hap K positive and 20% will not have the Hap K positive result.

All patients will be screened for eligibility based on the haplotype status. Patients will be randomized to either veliflapon or placebo on top of standard care. Patients are randomized within 5-30 days of their ACS event.

This is an events driven study with the time of the first occurrence of any of the following elements: hospitalization for UA or urgent revascularization, fatal/non-fatal MI, fatal/non-fatal stroke and CV related death comprising the primary endpoint. The primary null hypothesis of efficacy is that time to first CV event among African American patients with a positive LTA4H HapK Variant assay test is no different from placebo when either is given in addition to standard of care therapy. A total of 3450 eligible patients will be randomized in this study.

The treatment duration for patients enrolled in the study will be a target of at least 6 months (based on approximate time of last patient enrolled) and up to 36 months (from first patient enrolled). All cardiac clinical events endpoints will be adjudicated by an independent Clinical Endpoint Committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 35 years of age or older
* African American by self-report.
* A history of either acute MI or admission for unstable angina (UA)within 30 days of randomization
* Women who have undergone surgical sterilization (hysterectomy or bilateral tubal ligation or bilateral oophorectomy)or are > 2 years post-menopausal by medical history are also eligible.
* Women of childbearing potential must have a negative urine pregnancy test and are required to use 2 barrier methods of contraception throughout the study.
* Patients are capable of understanding study procedures and agree to participate in the study including scheduled follow up visits and consent to genetic haplotype testing.

Exclusion Criteria:

* Presence of active, symptomatic HF defined by presence of New York Heart Association Class II-IV at time of screening.
* Received any treatment with an investigational agent or device within 4 weeks.
* Evidence of secondary angina or ischemia
* Underlying cardiac disorders that may cause cardiac ischemia including aortic stenosis or hypertrophic cardiomyopathy.
* Presence of active hepatic disease or AST and/or ALT > 3.0 × ULN.
* Calculated creatinine clearance < 30 ml/minute OR the presence of chronic and severe renal insufficiency.
* Major surgery performed within six weeks prior to scheduled day of randomization.
* Any other major intercurrent illness and other condition, which, in the opinion of the Investigator, will interfere with the patient's participation in the study or leads to a survival prognosis of < 5 years.
* A history of additional risk factors for Torsades de Pointe (TdP)
* Patients who are not willing to return for follow up visits or with a known history of non-compliance.
* Patients who consume > 3 alcoholic drinks/day or > 15 drinks/week, or have a history of alcohol abuse within the past 2 years.
* History of active drug abuse within 1 year of screening for the study.
* Pregnant or lactating women.
* Poor mental function or any other reason that may cause difficulty in complying with the requirements of the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3450
Dates: Start 2006-05

PRIMARY OUTCOMES:
Time to first occurrence of a composite endpoint including:hospitalization for unstable angina or urgent revascularization; fatal/non-fatal MI; fatal/non-fatal stroke or CV related death

SECONDARY OUTCOMES:
Time to first occurrence of each of the following: an acute CV event (one of the composite CV events) among ALL randomized patients; MI, fatal and non-fatal
Stroke, fatal and non-fatal; CV related death and all cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Weaver, M.D., Principal Investigator — Henry Ford Hospital; Christopher Granger, M.D., Principal Investigator — Duke University
Locations (11):
- United States (11):
  - Montgomery, Alabama
  - Jacksonville, Florida
  - Melrose Park, Illinois
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Carrollton, Texas
  - Fort Worth, Texas
  - Richardson, Texas
  - Hopewell, Virginia
  - Suffolk, Virginia